CLINICAL TRIAL: NCT02025959
Title: Sleep for Inpatients: Empowering Staff to Act
Acronym: SIESTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-1766
Record Dates: First submitted 2013-12-17; First posted 2014-01-01 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Sleep Disorders; Sleep
Keywords: staff empowerment; Sleep Apnea; educational intervention
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Apnea Syndromes | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Educational Intervention (Experimental): Educating hospital staff on good sleep hygiene for patients and screening for sleep disorders
  Interventions: Behavioral: Educating hospital staff on good sleep hygiene for patients and screening for sleep disorders

INTERVENTIONS:
Behavioral: Educating hospital staff on good sleep hygiene for patients and screening for sleep disorders

SUMMARY:
Getting better sleep in the hospital is especially important due to a variety of adverse health effects that can potentially worsen patient recovery.

To address these concerns and improve sleep in US hospitals, we aim to develop the SIESTA (Sleep for Inpatients: Empowering Staff to Act) program as an educational intervention designed to prepare hospital staff to assist patients in obtaining better sleep in hospitals and recognize the importance of screening for sleep disorders. The major educational goals of this proposal is to develop and pilot test an online educational program (SIESTA) which aims to train and motivate medical professionals to provide better sleep for hospitalized patients.

We will utilize data from an ongoing sleep study, performed by the research team at the University of Chicago that looks at how adult patients are able to sleep while they are in the hospital, as a means of education for the participating medical staff.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, the subjects must be University of Chicago hospital employees over the age of 18 years old.

Exclusion Criteria:

* We will exclude any hospital staff under the age of 18 years old from this study as well as hospital patients and non-hospital staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-08; Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Impact of Educational program | Four years
  We will assess if the SIESTA program translates into behavior change based on staff satisfaction, knowledge, behavior and qualitative analysis.

SECONDARY OUTCOMES:
Patient Outcomes | Four Years
  We will asses affect of Intervention on hospitalized patient outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Vineet M Arora, MD, MAPP, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Result] Shear TC, Balachandran JS, Mokhlesi B, Spampinato LM, Knutson KL, Meltzer DO, Arora VM. Risk of sleep apnea in hospitalized older patients. J Clin Sleep Med. 2014 Oct 15;10(10):1061-6. doi: 10.5664/jcsm.4098. PMID 25317085